CLINICAL TRIAL: NCT04099459
Title: ORCA Study: Osteoarthritis and Risks Associated With the Consumption of NSAIDs
Acronym: ORCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Scandinavia Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: ORCA
Record Dates: First submitted 2019-09-16; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cross-sectional epidemiological study in patients with diagnosis of osteoarthritis (OA) in order to evaluate risk factors associated with the use / prescription of non-steroidal anti-inflammatory drugs (NSAID).

DETAILED DESCRIPTION:
OBJECTIVE: To evaluate the presence of risk factors associated with the use / prescription of non-steroidal anti-inflammatory drugs (NSAID) in patients diagnosed with osteoarthritis (OA).

MATERIALS AND METHODS: A multicentric, cross-sectional epidemiological study, will be carried out in patients ≥ 38 years of age, with a previous diagnosis of primary or secondary OA, according to criteria of the American College of Rheumatology (ACR). The presence of at least one risk factor for the use / prescription of NSAIDs is the main variable. The secondary variables to be evaluated include: Demographical characterization of the patients, current disease status (level of pain and functional limitation), treatment (s) used (related or not to OA) and events side effects associated with the treatment (s). The analysis will be carried out from two perspectives: A first descriptive approach and a second analytical approach.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 38 years
* Previous diagnosis of OSTEOARTRITIS (primary or secondary) at least 30 days before or more, in at least one or more of the following locations: Knee and / or Hip and / or Hand, according to criteria of the American College of Rheumatology (ACR)

Exclusion Criteria:

* Refusal to participate in the study by the patient.
* Patients who, in the judgment of the Investigator, do not understand or are not willing to adequately answer to the questions.
* Mental or psychiatric illness that, in the judgment of the investigator, does not allow adequate information to be obtained.

Min Age: 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colombian patients, ≥ 38 years, with previous diagnoses of OSTEOARTRITIS.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Presence of risk factors for adverse events associated to consumption of NSAIDs | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years
  A descriptive analysis about presence of risk factors for the possible ocurrence of adverse events associated to consumption of NSAIDs in the patients: gastrointestinal, renal, cardiovascular.

SECONDARY OUTCOMES:
Demographic analysis | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years
  Characterization of patients
List of drugs used (by the patient) for treatment of osteoarthritis (OA) | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years
  List of drugs used (by the patient) for treatment of osteoarthritis (OA), including time of use and posology.
Evaluation of the current state of the disease according to functional limitation and pain | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years
  Evaluation of functional limitation and pain according to the Visual Analogue Scale graduated between 0 and 10, being 0 absence or asymptomatic and 10 the maximum pain or maximum functional limitation.
Adverse Events related with the treatments | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years
  Evaluation of Adverse events associated with the treatment (s)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Castillo, Dr, Study Director — Medical Director
Locations (1):
- Scandinavia Pharma, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No